CLINICAL TRIAL: NCT04865744
Title: The Effect of Semaglutide on Pituitary Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tartu (Other)
Responsible Party: Principal Investigator, Vallo Volke, Professor, University of Tartu
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: Sema21
Record Dates: First submitted 2021-04-28; First posted 2021-04-29 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — semaglutide; Tablets

STUDY DESIGN:
Intervention Model Description: Blinded Randomised Single-group Crossover
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oral semaglutide 7 mg (Active Comparator): The semaglutide 7 mg tablet taken orally with upto120 ml of water.
  Interventions: Drug: Semaglutide 7 MG Oral Tablet
- Placebo (Placebo Comparator): The placebo tablet taken orally with 120 ml of water.
  Interventions: Drug: Placebo
- Oral semaglutide 14 mg (Active Comparator): The semaglutide 14 mg tablet taken with upto 120 ml of water.
  Interventions: Drug: Semaglutide 14 MG Oral Tablet

INTERVENTIONS:
Drug: Semaglutide 7 MG Oral Tablet — Semaglutide 7 mg oral tablet taken after an overnight fast with up to 120 ml of water.
  Other Names: Rybelsus 7 mg
  Arms: Oral semaglutide 7 mg
Drug: Placebo — Placebo tablet is taken after an overnight fast with up to120 ml of water.
  Arms: Placebo
Drug: Semaglutide 14 MG Oral Tablet — Semaglutide 14 mg oral tablet taken after an overnight fast with up to 120 ml water.
  Other Names: Rybelsus 14 mg
  Arms: Oral semaglutide 14 mg

SUMMARY:
The primary aim of the study is to describe the effect of a single oral dose of semaglutide 7 mg on growth hormone secretion.

DETAILED DESCRIPTION:
The randomized blinded placebo-controlled clinical trial is conducted on 10 healthy volunteers.

5 study subjects receive once 7 mg of oral semaglutide and once placebo. 5 study subjects receive once 14 mg of oral semaglutide and once placebo. The study group and order of administration of study medication are decided on randomization. The placebo and oral semaglutide are administered at least 4 weeks apart.

Blood samples are taken before and during 4 hours after the study medication administration (at 60, 90, 120, 150, 180, and 240 minutes after study medication administration).

The primary endpoint is the peak value of growth hormone measured during the 4 hours after study medication administration.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* The body weight >65 kg

Exclusion Criteria:

* presence of chronic illness
* the daily use of medications
* pregnancy
* lactation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2021-05-19 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Growth hormone peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration.

SECONDARY OUTCOMES:
Cortisol peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration.
Adrenocorticotropin (ACTH) peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration.
Aldosterone peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration.
Glucose nadir | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Lowest glucose concentration measured after study medication administration
C-peptide peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration.
Copeptin peak | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  Maximum concentration measured after study medication administration

OTHER OUTCOMES:
Nausea | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  The intensity of nausea on a 0-10 points visual analog scale, where 0 indicates no nausea and 10 worst imaginable nausea.
Heart rate | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  The change in heart rate compared to baseline
Blood pressure | 60, 90, 120, 150, 180 and 240 minutes after study medication administration
  The change in blood pressure compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Vallo Volke, MD, PhD, Principal Investigator — University of Tartu
Locations (1):
- Tartu University Hospital, Tartu, Estonia

IPD SHARING:
Plan to Share IPD: No